CLINICAL TRIAL: NCT02176187
Title: A Randomised Open Label, Four Way, Cross-over Scintigraphic Evaluation of the Respimat® Inhaler vs a Metered Dose Inhaler (HFA-MDI) Using Berodual® in Patients With Chronic Obstructive Pulmonary Disease (COPD) With Poor MDI Technique
Brief Title: Berodual® Respimat® vs Metered Dose Inhaler in Patients With Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 215.1360
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (2):
- natural technique, without instructions (Experimental): randomised sequence of Berodual® Respimat® and Berodual® MDI
  Interventions: Drug: Berodual® Respimat® inhaler; Drug: Berodual® metered dose inhaler
- optimal technique, with instructions (Experimental): randomised sequence of Berodual® Respimat® and Berodual® MDI
  Interventions: Drug: Berodual® Respimat® inhaler; Drug: Berodual® metered dose inhaler

INTERVENTIONS:
Drug: Berodual® Respimat® inhaler — fenoterol hydrobromide 50μg + ipratropium bromide 20μg
Drug: Berodual® metered dose inhaler — fenoterol hydrobromide 50μg + ipratropium bromide 20μg

SUMMARY:
Study to compare the effect of 'natural' as opposed to 'optimal' technique on the percentage of the dose received from the Respimat® inhaler and metered dose inhaler

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of COPD and must meet the following spirometric criteria:

  * Patients must have relatively stable, mild to severe airway obstruction with an forced expiratory volulme in one second (FEV1) ≤70% of predicted normal and FEV1 ≤70% of forced vital capacity (FVC). Predicted normal values calculated according to evolutionary conserved chromosome segments (ECCS)
  * Patients who have frequent exacerbations which could be expected to interfere with the patient's ability to participate in the study should be excluded
* Male or non-pregnant/non-lactating female patients aged ≥18 years
* Patients must demonstrate poor MDI technique prior to the start of the study. Presence of any of the following will be considered poor technique:

  * Failure to co-ordinate "firing" of an MDI with inhalation
  * Too fast an inhalation rate (> 30 litres/minute (L/min))
  * Presence of "Cold Freon" effect (MDI spray hitting the back of the throat that caused the patient to stop inhaling)
* All patients must sign an informed consent form prior to participation in the study, i.e. prior to pre-study washout of their usual pulmonary medications
* Current or ex-smokers with a smoking history of >10 pack years

Exclusion Criteria:

* Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
* Patients with clinically relevant abnormal baseline haematology, blood chemistry or urinalysis, if the abnormality defines a disease listed as an exclusion criterion will be excluded
* Patients with a recent history (i.e. six months or less) of myocardial infarction
* Patients with any unstable or life-threatening cardiac arrhythmia or who have been hospitalised for heart failure within the past year
* Patients who regularly use daytime oxygen therapy for more than 1 hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen
* Patients with known active tuberculosis
* Patients with a history of cancer within the last five years. Patients with treated basal cell carcinoma are allowed
* Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis
* Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion 1
* Patients with any upper respiratory infection in the past 14 days prior to the screening visit or during the baseline period
* Patients who are currently in a pulmonary rehabilitation programme or who have completed a pulmonary rehabilitation programme in the six weeks prior to the screening visit
* Patients with known hypersensitivity to β2-agonists, anticholinergic drugs or any excipients of the active or placebo Berodual®
* Patients with known narrow-angle glaucoma
* Patients who are being treated with antihistamines (H1 receptor antagonists)
* Patients using oral corticosteroid medication at unstable doses (i.e. less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisolone per day or 20 mg every other day
* Patients who are being treated with monamine oxidase inhibitors or tricyclic antidepressants
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e. oral or injectable eg Depo-Provera or Noristerat contraceptives, intrauterine devices, diaphragm (plus spermicide) or subdermal implants eg: Norplant®)
* Patients with, in the opinion of the investigator, a history of and/or active significant alcohol or drug abuse
* Patients who have taken an investigational drug within four months or six half lives (whichever is the greater) prior to screening visit and/or the administration of radiolabelled dosage forms within the three months prior to the screening visit
* Radiation exposure from clinical studies, including that from the present study and diagnostic X-rays but excluding background radiation, exceeding 5 millisievert (mSv) in the last 12 months or 10 mSv in the last five years. No patient whose occupational exposure is monitored will participate in the study

Precautions: As with other anticholinergic drugs, Berodual® should be used with caution in patients with prostatic hyperplasia or bladder neck obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2003-04; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Percentage of dose in the whole lung | immediately after dosing
  Deposition of aerosol via gamma scintigraphy

SECONDARY OUTCOMES:
Percentage of dose in the central lung zone | immediately after dosing
  Deposition of aerosol via gamma scintigraphy
Percentage of dose in the intermediate lung zone deposition | immediately after dosing
  Deposition of aerosol via gamma scintigraphy
Percentage of dose in the peripheral lung zone deposition | immediately after dosing
  Deposition of aerosol via gamma scintigraphy
Peripheral lung zone/central lung zone deposition ratio (lung penetration index) | immediately after dosing
  Deposition of aerosol via gamma scintigraphy
Percentage of dose in oropharyngeal deposition | immediately after dosing
  Deposition of aerosol via gamma scintigraphy